CLINICAL TRIAL: NCT06053528
Title: Pattern and Outcome of Respiratory Diseases in Patients Admitted in the Chest Department at Assiut University Hospital
Brief Title: Pattern and Outcomes of Chest Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Hamdan Zaki Adeel, Resident doctor, Assiut University
Other Study IDs: Pattern of chest diseases
Record Dates: First submitted 2023-09-01; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Chest--Diseases
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antibiotic — Effect if treatment

SUMMARY:
The objective of this study is to determine the pattern and outcome of respiratory diseases in adults patients admitted to the Department of Chest Diseases at Assiut University Hospital.

DETAILED DESCRIPTION:
Respiratory diseases constitute an important global health burden. Pneumonia, tuberculosis, obstructive and restrictive lung diseases, pleural diseases, and malignancies are common respiratory conditions for hospital admission.Before the emergence of COVID-19, pneumonia, including community-acquired pneumonia (CAP) and hospital-acquired pneumonia (HAP)/ventilation-associated pneumonia (VAP), was one of the most common infectious diseases, and could cause major health problems, associated with high morbidity and mortality in all age groups worldwide . The outbreak of COVID-19 has significantly changed the epidemiology of respiratory tract infection. More than 376 million people have been infected and 5 million have died in the whole world. This in addition to the long term post COVID pulmonary sequelae. Chronic obstructive pulmonary disease (COPD), lower respiratory tract infections, lung cancer and tuberculosis have been identified as top four respiratory diseases among ten leading causes of death worldwide. The forum of international respiratory societies (FIRS) estimated that 65 million people have moderate to severe COPD resulting in 3 million deaths per year, making it third leading cause of death worldwide .Currently, asthma affects an estimated 334 million people worldwide and is projected to increase to 400 million by the year 2025 .

In ;2015 10,4million people developed TB with 1.4 million global deaths were reported.

Neoplasms of the lungs are the leading cause of cancer incidence and mortality worldwide.

ELIGIBILITY:
Inclusion Criteria:

* All adults patients admitted to the Chest Department during the study period will be included.

Exclusion Criteria:

* Patients who will die, be discharged, or be transferred before completing data collection will be excluded from our study.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Prospective, descriptive and analytical study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Determine number of patients who experience improvement on discharge | One year
Number of patient who Transferred to another hospital forcontintreatment | One year
Number of patient died while on admission | One year
Number of patient who Discharged against medical advice | One year

REFERENCES:
- See also: Global Asthma Report [Internet]. Auckland: Global Asthma Network; 2014. Available from — http://globalasthmanetwork.org/publications/Global_Asthma_Report_2014.pdf